CLINICAL TRIAL: NCT05715385
Title: Comparison Between Grid Macular Laser and Topical Bromfenac 0.09% in the Treatment of Diabetic Macular Edema
Brief Title: Comparison of Treatments in Diabetic Macular Edema
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Babasaheb Ambedkar Memorial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 226-31122-142-201800
Record Dates: First submitted 2023-01-13; First posted 2023-02-08 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Laser photocoagulation (Active Comparator): Grid laser was performed under topical anesthesia with frequency doubled Nd YAG laser of wavelength 532 nm.
  Laser Parameters for grid photocoagulation Lens used: Mainster grid lens Spot size: 75-100μ The burn intensity for grid laser: barely visible (light grey) Power: 80-100mw depending on the condition of the laser, the opacities in the media and background pigmentation.
  Duration: 100msec No. of spots: 80-100 Laser burns were placed at least one burn width apart. Wider if the thickening was less severe. If necessary, the grid laser extended up to 2 disc diameters superiorly, inferiorly and temporally from the centre of the macula. Treating the area within 500 microns of the disc margin or the centre of the macula was avoided.
  Interventions: Procedure: laser photocoagulation
- Bromfenac 0.09% (Active Comparator): Twice daily eye drop bromfenac 0.09% for 6 weeks
  Interventions: Drug: eye drop bromfenac 0.09%
- Observation (Placebo Comparator): Eye drop carboxymethyl cellulose 0.5% to be instilled thrice a day for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Procedure: laser photocoagulation — Laser Parameters of grid photocoagulation Diffuse diabetic macular edema is treated by a grid pattern of laser. The grid is applied to areas of retinal thickening with diffuse leakage or capillary non-perfusion.
  Spot size: 50-100 micron is utilized. The burn intensity for grid laser: barely visible (light grey). Power of laser burn is between 80-100 mw depending on the condition of the laser, the opacities in the media and background pigmentation.
  Laser burns should be placed at least one burn width apart, wider if thickening is less severe. If necessary, the grid can extend up to 2 disc diameters superiorly, inferiorly, and temporally from the centre of the macula. One should avoid treating within 500 microns of the disc margin or the centre of the macula.
  Duration of about 0.05-0.1 sec is used Number of spots- 100-500
  Arms: Laser photocoagulation
Drug: eye drop bromfenac 0.09% — twice daily e/d bromfenac 0.09% for 6 weeks
  Arms: Bromfenac 0.09%
Drug: Placebo — Observation group. No intervention done. Only eye drop carboxymethyl cellulose 0.5% to be instilled thrice a day for 6 weeks.
  Arms: Observation

SUMMARY:
Prospective or cohort study to compare the effects of grid macular laser, topical bromfenac 0.09% and placebo (carboxymethyl cellulose 0.5%) medication in diabetic macular edema.

60 eyes with macular edema of two types i.e. cystoid macular edema (CME) and clinically significant macular edema (CSME) were divided into three groups with 20 patients in each group. One group was treated with grid laser photocoagulation, the second group was treated with topical bromfenac 0.09% drops two times a day and the third group was treated with topical carboxy methyl cellulose 0.5% three times a day (placebo treatment).

DETAILED DESCRIPTION:
Study site:

Dr Babasaheb Ambedkar Memorial Hospital, of the Central Railway at Byculla, Mumbai.

Study Population:

Patients attending Ophthalmology Out Patient Department(OPD) at Dr Babasaheb Ambedkar Memorial Central Railway Hospital, Byculla, Mumbai.

Study design:

Prospective or cohort study to compare the effects of grid macular laser, topical bromfenac 0.09% and placebo (carboxymethyl cellulose 0.5%) medication in diabetic macular edema.

Sample size with justification:

60 eyes fulfilling the selection criteria were included in the study after informed consent.

Justification of sample size:

To calculate sample size formula used is N = Z2 * P (1-P) D2 Where, Z = standard normal deviate =1.96 (at 95% confidence interval) D = margin of error (precision) will be 0.05 P = Prevalence. According to Chennai Epidemiological Study99, the prevalence of diabetic retinopathy in India is 17.6%. Out of these, less than one third patients have mild macular edema.

So calculated sample size is 60 patients.

Time frame of the study:

Patients were randomly selected from those who were attending the OPD from November 2014 to October 2015.

Sampling procedure and data collection:

All the patients enrolled in the study were informed verbally about potential benefits and risks associated with the treatment modalities and a fully informed written consent was obtained from each of them.

A detailed history was obtained in each case. A thorough ophthalmic history regarding mode of onset of symptoms, duration of symptoms, a history of any previous intervention in the affected eye, medical history including duration of diabetes mellitus, medications being taken, and history of any other systemic illness was obtained and recorded on case record sheet. A comprehensive ophthalmic examination of all patients was done.

The patients were then divided by simple random sampling into three groups. One group was treated with grid laser photocoagulation, the second group was treated with topical bromfenac 0.09% drops two times a day and the third group was treated with topical carboxy methyl cellulose 0.5% three times a day (placebo treatment).

HISTORY AND EXAMINATION INCLUDED:

i. General information: Name, age and sex ii. Chief complaints: The complaints patient presented with along with its onset, duration and progress.

iii. Ophthalmic history:

* History of any ocular disease or injury which may affect vision and treatment taken for it.
* History of undergoing any ocular procedure. iv. History of diabetes mellitus especially with regard to its duration and treatment v. Visual acuity: Best corrected visual acuity (BCVA) testing was done on the ETDRS chart and values were obtained in logMAR for analysis.

vi. Intraocular pressure measurement: Measured using Goldman applanation tonometer under topical anesthesia. vii. Slit lamp examination: For anterior segment examination to ensure clarity of lens and cornea.

viii. Fundus examination: Fundus examination was done with slit lamp biomicroscopy using 60 dioptre lens and indirect ophthalmoscopy. Photographs were taken with fundus camera.

ix. Optical coherence tomography (OCT) It was done at the beginning of the study before doing any intervention and then again after 6 weeks.

PROCEDURE:

* OCT machine used was Spectral Domain Cirrhus OCT from Carl Zeiss (Cirrhus High Definition-OCT)
* The pupils were dilated and the patient was positioned at the machine.
* A 512 * 128 macular cube protocol was chosen, consisting of 128 horizontal scan lines, each consisting of 512 A-scans per line. The instrument provided a retinal thickness map: 3 concentric circular areas were centered on the fixation point. The diameter of each was 1, 3 and 6 mm. In each one of these 9 areas, the software calculated the mean value from all the thickness measurements on each single A-scan. In addition to average retinal thickness of 9 zones, including a 1 mm central zone, the Cirrus macula readout provided macular volume and average macular thickness, which reflected the 3D structure of retina.
* The retinal thickness was measured from retinal pigment epithelium (RPE) to internal limiting membrane (ILM).
* Central macular thickness was calculated as mean thickness in the central 1000 um diameter area.

  x. Blood Investigations: Blood was checked for fasting blood sugar, post prandial blood sugar and HbA1c levels. The blood tests were repeated at the end of 6 weeks.

PROCEDURE OF GRID PHOTOCOAGULATION For the patients treated with laser photocoagulation, grid laser was performed under topical anesthesia with frequency doubled neodymium-doped yttrium aluminum garnet (Nd YAG) laser of wavelength 532 nm.

Laser Parameters for grid photocoagulation Lens used: Mainster grid lens Spot size: 75-100μ The burn intensity for grid laser: barely visible (light grey) Power: 80-100mw depending on the condition of the laser, the opacities in the media and background pigmentation.

Duration: 100msec No. of spots: 80-100 Laser burns were placed at least one burn width apart. Wider if the thickening was less severe. If necessary, the grid laser extended up to 2 disc diameters superiorly, inferiorly and temporally from the centre of the macula. Treating the area within 500 microns of the disc margin or the centre of the macula was avoided.

Patients in the bromfenac group were given twice daily e/d bromfenac 0.09% for 6 weeks.

Patients in the placebo group were given e/d carboxymethyl cellulose 0.5% to be instilled thrice a day for 6 weeks.

Follow up The patients were called every week and their visual acuity and fundus was checked.

The patients were instructed to maintain a good control diabetes, blood pressure and adhere to their follow up regimen and to report at the first sign of worsening vision.

The visual acuity, fundus photograph, macular thickness on OCT at 6 weeks checkup were used in present analysis.

Ethical consideration:

The investigator sought ethical clearance from Dr Babasaheb Ambedkar Memorial Central Railway Hospital, Byculla, Mumbai, ethical and scientific committee. Patients were included in this study only after they gave informed consent. Patients were informed of the purpose of the study, procedures to be performed and the risks and benefits of the treatment. As patients were on regular weekly follow up where vision and fundus was checked, even those patients receiving placebo had the benefit of a careful monitoring in place for intervention if required.

Data Management and Statistical Analysis:

* After data collection, data entry was done in excel.
* Statistical analysis was performed with the help of the software SPSS ver 15.
* For comparing quantitative data

  * Between the study groups chi square test was applied
  * Within the group that is before and after the study, paired 't' test was applied
* Comparison of non- parametric (qualitative) data between the study groups was done using Fisher Exact test
* Statistical significance is indicated by conventional symbols:

  * p <0.05: Statistically significant

    * p >0.05: Statistically non-significant

ELIGIBILITY:
Inclusion Criteria:

* Patient with type 1 or type 2 diabetes.
* The study eye met the following:

  * OCT thickness of the macula upto 400 microns.
  * On clinical examination, definite retinal thickening due to diabetic macular edema within 3000 μm of the center of the macula.
* Patient with well controlled blood sugar levels i.e. fasting blood sugar level < 110mg% and post prandial blood sugar level < 126 mg%. Also HbA1c level less than 7%.
* Able and willing to provide informed consent.
* Media clarity, pupillary dilation, and study participant cooperation sufficient for adequate OCT and fundus photographs.
* Normal optic disc.

Exclusion Criteria:

* Use of systemic corticosteroids for any other systemic condition or previous anti-Vascular endothelial growth factor (VEGF) therapy.
* Current use of prescription systemic NSAIDs.
* Known allergy to bromfenac.
* History of use of NSAID eye drops within the last 30 days or anticipated need for such drops during the study due to other ocular conditions.
* Any ocular condition, coexisting with diabetic macular edema, which might affect visual acuity.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in visual acuity in laser photocoagulation group | Baseline and 6 weeks
  Best corrected visual acuity will be measured by logMAR scale
Change in visual acuity in bromfenac group | Baseline and 6 weeks
  Best corrected visual acuity will be measured by logMAR scale
Change in visual acuity in observation group | Baseline and 6 weeks
  Best corrected visual acuity will be measured by logMAR scale

OTHER OUTCOMES:
Change in central macular thickness in laser photocoagulation group | Baseline and 6 weeks
  Central macular thickness measured by OCT
Change in central macular thickness in bromfenac group | Baseline and 6 weeks
  Central macular thickness measured by OCT
Change in central macular thickness in observation group | Baseline and 6 weeks
  Central macular thickness measured by OCT

CONTACTS AND LOCATIONS:
Overall Officials: Mehul Joshi, FRCS,DNB, Principal Investigator — Dr Babasaheb Ambedkar Central Railway Hospital, Byculla, Mumbai, Maharashtra, India; Arundhati Malviya, MS(Ophthal), Study Chair — Dr Babasaheb Ambedkar Central Railway Hospital, Byculla, Mumbai, Maharashtra, India; Memuna Bahadur, MS(Ophthal), Study Chair — Dr Babasaheb Ambedkar Central Railway Hospital, Byculla, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and findings will be made available as open source for all other researchers.
Supporting Information: Study Protocol
Time Frame: The data will be submitted for publication in the Indian Journal of Ophthalmology after approval by the clinicialtrials.gov registration department and will be available there always for reference.
Access Criteria: Keywords to access the study will be Diabetic macular edema; Bromfenac; Laser photocoagulation

REFERENCES:
- [Background] Pinna A, Blasetti F, Ricci GD, Boscia F. Bromfenac eyedrops in the treatment of diabetic macular edema: a pilot study. Eur J Ophthalmol. 2017 May 11;27(3):326-330. doi: 10.5301/ejo.5000888. Epub 2016 Nov 16. PMID 28009414
- [Background] Busch C, Fraser-Bell S, Zur D, Rodriguez-Valdes PJ, Cebeci Z, Lupidi M, Fung AT, Gabrielle PH, Giancipoli E, Chaikitmongkol V, Okada M, Lains I, Santos AR, Kunavisarut P, Sala-Puigdollers A, Chhablani J, Ozimek M, Hilely A, Unterlauft JD, Loewenstein A, Iglicki M, Rehak M; International Retina Group. Real-world outcomes of observation and treatment in diabetic macular edema with very good visual acuity: the OBTAIN study. Acta Diabetol. 2019 Jul;56(7):777-784. doi: 10.1007/s00592-019-01310-z. Epub 2019 Mar 22. PMID 30903434
- [Background] Baklayan GA, Munoz M. The ocular distribution of (14)C-labeled bromfenac ophthalmic solution 0.07% in a rabbit model. Clin Ophthalmol. 2014 Sep 4;8:1717-24. doi: 10.2147/OPTH.S66638. eCollection 2014. PMID 25228788
- [Background] Schoenberger SD, Kim SJ. Nonsteroidal anti-inflammatory drugs for retinal disease. Int J Inflam. 2013;2013:281981. doi: 10.1155/2013/281981. Epub 2013 Jan 14. PMID 23365785
- [Background] Waterbury LD, Silliman D, Jolas T. Comparison of cyclooxygenase inhibitory activity and ocular anti-inflammatory effects of ketorolac tromethamine and bromfenac sodium. Curr Med Res Opin. 2006 Jun;22(6):1133-40. doi: 10.1185/030079906X112471. PMID 16846546
- [Background] Ahmadi MA, Lim JI. Update on laser treatment of diabetic macular edema. Int Ophthalmol Clin. 2009 Spring;49(2):87-94. doi: 10.1097/IIO.0b013e31819fd6b2. No abstract available. PMID 19349789